CLINICAL TRIAL: NCT01255410
Title: A Phase I Study of the Safety and Immunogenicity of the Recombinant Live-Attenuated Human Metapneumovirus Vaccine, rHMPV-Pa Lot HMPV #101A, Delivered as Nose Drops to Adults 18 to 49 Years of Age, HMPV-Seropositive Children 12 to 59 Months of Age, and HMPV-Seronegative Infants and Children 6 to 59 Months of Age
Brief Title: Evaluation of the Safety and Immunogenicity of a Live Attenuated Human Metapneumovirus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIR 271
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Metapneumovirus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Healthy Adults (Group 1) (Experimental): Healthy adults will receive a single dose of 10^6 plaque forming unit (PFU) rHMPV-Pa vaccine intranasally.
  Interventions: Biological: 10^6 PFU rHMPV-Pa vaccine
- Seropositive Children-Vaccine (Group 2) (Experimental): Seropositive children will receive a single dose of 10^6 PFU rHMPV-Pa vaccine intranasally.
  Interventions: Biological: 10^6 PFU rHMPV-Pa vaccine
- Seropositive Children-Placebo (Group 2) (Placebo Comparator): Seropositive children will receive a single dose of placebo vaccine intranasally.
  Interventions: Biological: Placebo Vaccine
- Seronegative Infants and Children-Vaccine (10^5) (Group 3) (Experimental): Seronegative infants and children will receive a single dose of 10^5 PFU rHMPV-Pa vaccine intranasally.
  Interventions: Biological: 10^5 PFU rHMPV-Pa vaccine
- Seronegative Infants and Children-Placebo (Group 3) (Placebo Comparator): Seronegative infants and children will receive a single dose of placebo vaccine intranasally.
  Interventions: Biological: Placebo Vaccine
- Seronegative Infants and Children-Vaccine (10^6) (Group 4) (Experimental): Seronegative infants and children will receive a single dose of 10^6 PFU rHMPV-Pa vaccine intranasally.
  Interventions: Biological: 10^6 PFU rHMPV-Pa vaccine
- Seronegative Infants and Children-Placebo (Group 4) (Placebo Comparator): Seronegative infants and children will receive a single dose of placebo vaccine intranasally.
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: 10^6 PFU rHMPV-Pa vaccine — Single dose of 10^6 PFU rHMPV-Pa vaccine delivered intranasally
  Arms: Healthy Adults (Group 1); Seronegative Infants and Children-Vaccine (10^6) (Group 4); Seropositive Children-Vaccine (Group 2)
Biological: 10^5 PFU rHMPV-Pa vaccine — Single dose of 10^5 PFU rHMPV-Pa vaccine delivered intranasally
  Arms: Seronegative Infants and Children-Vaccine (10^5) (Group 3)
Biological: Placebo Vaccine — Single dose of placebo vaccine delivered intranasally
  Arms: Seronegative Infants and Children-Placebo (Group 3); Seronegative Infants and Children-Placebo (Group 4); Seropositive Children-Placebo (Group 2)

SUMMARY:
People who are infected with human metapneumovirus (HMPV) may develop upper and lower respiratory illnesses. Children are particularly sensitive to HMPV infection. This study will evaluate the safety and immune response of an HMPV vaccine in healthy adults, HMPV-seropositive children, and HMPV-seronegative infants and children.

DETAILED DESCRIPTION:
HMPV is a viral respiratory pathogen that was discovered in 2001, but studies have shown that it has been circulating in humans for at least 50 years. Older adults and adults with asthma who are infected with HMPV may be at increased risk for lower respiratory illness and hospitalization. In infants and young children, HMPV infection may cause upper or lower respiratory illness, ear infections, bronchiolitis, croup, pneumonia, and exacerbations of asthma. Children less than 2 years of age are most susceptible to severe HMPV infections, and HMPV is the second or third leading cause of viral lower respiratory illness in children. The National Institute of Allergy and Infectious Diseases (NIAID) is working to develop a live-attenuated, intranasally administered HMPV vaccine for use in infants. The purpose of this study is to evaluate the safety and immunogenicity of an HMPV vaccine.

The vaccine will be evaluated in four groups of participants: healthy adults; HMPV-seropositive children; and two groups of HMPV-seronegative infants and children, with each seronegative group receiving a different dose of the vaccine. In the adult group, participants will all receive the vaccine; in the infant and children groups, participants will be randomly assigned to receive either the vaccine or a placebo. Study researchers will review participants' study data and confirm the safety of the vaccine before enrolling the next group of participants.

This study will first enroll healthy adults. At a baseline study visit, all participants will undergo a medical history review, physical examination, nasal wash procedure, vital sign measurements, and a blood collection. They will then receive the vaccine, and they will remain in the clinic for 30 minutes for observation. Participants will record their temperature daily for 12 days. Additional study visits will occur at Days 3, 4, 5, 6, 7, 10, and 12. At each study visit, participants will undergo a medical history review, vital sign measurements, and a nasal wash procedure. A final study visit will occur on Day 28 and will also include a blood collection. The second group of participants will include seropositive children. They will receive the vaccine or a placebo vaccine and take part in the same study procedures as the adult participants. Participants' parents will receive telephone calls or e-mails from study staff on Days 1, 2, 8, 9, 11, and 13 to obtain and record medical history and temperature readings. The third and fourth groups of participants will include seronegative infants and children. Each of these two groups will receive different doses of the vaccine or placebo vaccine. They will attend study visits on Days 3, 5, 7, 10, 12, 14, 17, 19, 21, 28, and 56, and they will undergo the same study procedures as the other participants. Parents of seronegative infants and children will receive telephone calls or e-mails from study staff on Days 1, 2, 4, 6, 8, 9, 11, 13, 15, 16, 18, 20, 22 to 27, and 29.

Study staff will call all participants at Month 6 for a medical history review and follow up.

ELIGIBILITY:
Inclusion Criteria for Adults:

* Adult males and non-pregnant, non-nursing females 18 to 49 years old
* In good health without significant medical illness, physical examination findings, or significant laboratory abnormalities in urinalysis, complete blood count (CBC), alanine aminotransferase (ALT), or creatinine as determined by the investigator
* Available for the duration of the study
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must have negative urine pregnancy tests and must agree to use effective birth control methods (e.g., birth control pills, diaphragm and foam, condoms with spermicide, Depo-Provera) until 28 days after vaccination

Exclusion Criteria for Adults:

* Pregnant, as determined by a positive urine beta-human chorionic gonadotropin (HCG) test
* Breastfeeding
* Females of childbearing potential who are unwilling to practice effective birth control as described in the inclusion criteria
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the participant to understand and cooperate with the study protocol
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a participant in the study or would render the participant unable to comply with the protocol
* Has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the 12 months before study entry
* History of a severe allergic reaction or anaphylaxis
* History of splenectomy
* Current diagnosis of asthma in the 2 years prior to study entry
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory Western blot tests for HIV-1
* Positive ELISA and confirmatory immunoblot tests for hepatitis C (HCV)
* Positive ELISA HBsAg
* Abnormal urinalysis/urine dip
* Known immunodeficiency syndrome
* Current use of nasal or systemic steroid medications
* Receipt of blood products (including immunoglobulin) in the 3 months before study entry
* Current smoker unwilling to stop smoking for the duration of the study. More information on this criterion can be found in the protocol.
* Receipt of another investigational vaccine or investigational drug within 28 days of receiving this investigational HMPV vaccine
* Receipt of a live vaccine in the 4 weeks before study entry, a killed vaccine in the 2 weeks before study entry, or immune globulin within the 3 months prior to receiving the investigational vaccine
* Previous enrollment in an HMPV vaccine or viral challenge study
* Known hypersensitivity to any vaccine component
* Adults whose professional and/or personal responsibilities involve caring for children less than 59 months of age or for immunosuppressed individuals
* Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Body mass index (BMI) greater than 35

Inclusion Criteria for Seropositive Children:

* Healthy children 12 to 59 months of age, whose parent/guardian understands and signs the informed consent and who agrees to vaccine administration following a detailed explanation of the study
* Seropositive for HMPV as defined by serum neutralizing antibody titer greater than or equal to 1:40. If a child between 12 and 59 months of age is determined to be HMPV seropositive prior to Day 56, s/he does not need an additional screening serum specimen, but a prevaccination serum specimen must be obtained.
* Participant's history has been reviewed and they have undergone a physical examination indicating that s/he is in good health
* Available for the duration of the study

Exclusion Criteria for Seropositive Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy including systemic corticosteroids, or bone marrow/solid organ transplant recipients (topical steroids, topical antibiotics, and topical antifungal medications are acceptable)
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an HMPV vaccine
* Current use of nasal or systemic steroid medications
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. People with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. People who wheezed once or received bronchodilator therapy once in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months before study entry may also be enrolled.
* Member of a household that includes an immunocompromised individual or infants less than 12 months of age, other than a study participant
* Attends day care with infants less than 12 months of age, or immunosuppressed individuals, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.
* Receipt of another investigational vaccine or investigational drug within 28 days of receiving this investigational HMPV vaccine

Inclusion Criteria for Seronegative Infants and Children:

* Healthy children 6 to 59 months of age whose parents/guardians can understand and sign the informed consent and who agree to vaccine administration following detailed explanation of the study
* Seronegative for HMPV antibody as defined by serum neutralizing antibody titer less than 1:40 as determined within 42 days prior to inoculation
* Participant's history has been reviewed and they have undergone a physical examination indicating that s/he is in good health
* Available for the duration of the study

Exclusion Criteria for Seronegative Infants and Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy including systemic corticosteroids, or bone marrow/solid organ transplant recipients (topical steroids, topical antibiotics, and topical antifungal medications are acceptable)
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an HMPV vaccine
* Current use of nasal or systemic steroid medications
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. People with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. People who wheezed once or received bronchodilator therapy once in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months before study entry may also be enrolled.
* Member of a household that includes an immunocompromised individual or infants less than 12 months of age, other than a study participant
* Attends day care with infants less than 12 months of age and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.
* Receipt of another investigational vaccine or investigational drug within 28 days of receiving this investigational HMPV vaccine

Temporary Exclusion Criteria for All Age Groups:

The following are temporary or self-limiting conditions, and once resolved, the person may be enrolled, if otherwise eligible. If the period of temporary exclusion is more than 56 days for adults or HMPV-seropositive children, or more than 42 days for HMPV-seronegative children, participants will need to be rescreened.

* Fever (adult oral temperature of greater than or equal to 100.4°F [38°C], or pediatric rectal temperature of greater than or equal to 100.4°F [38.0°C]), acute upper respiratory illness (including nasal congestion significant enough to interfere with successful vaccination), or acute otitis media
* Received any killed vaccine or live attenuated rotavirus vaccine within the 2 weeks before study entry, any other live vaccine within the 4 weeks before study entry, or gamma globulin (or other antibody products) within the 3 months before study entry
* Received antibiotics or systemic or nasal steroid therapy for acute illness within the previous 3 days prior to vaccination (topical steroids and topical antibiotics or antifungal preparations are permitted)
* Infant or child participant has received salicylate (aspirin) or salicylate-containing products within the 1 month before study entry
* Children born at less than 37 weeks gestation will be deferred from participation until they are at least 1 year of age

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events that occur during the acute monitoring phase of the study | Measured at Days 0-12 for adult and seropositive participants, Days 0-28 for seronegative participants
Proportion of participants that develop 4-fold or greater rises in human metapneumovirus (HMPV) neutralizing antibody titer following vaccination. | Measured following the vaccination

SECONDARY OUTCOMES:
The number of vaccinated children and infants infected with rHMPV-Pa | Measured at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Janet Englund, MD, Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Herfst S, Fouchier RA. Vaccination approaches to combat human metapneumovirus lower respiratory tract infections. J Clin Virol. 2008 Jan;41(1):49-52. doi: 10.1016/j.jcv.2007.10.022. Epub 2007 Dec 4. PMID 18054841
- [Background] Williams JV, Harris PA, Tollefson SJ, Halburnt-Rush LL, Pingsterhaus JM, Edwards KM, Wright PF, Crowe JE Jr. Human metapneumovirus and lower respiratory tract disease in otherwise healthy infants and children. N Engl J Med. 2004 Jan 29;350(5):443-50. doi: 10.1056/NEJMoa025472. PMID 14749452